CLINICAL TRIAL: NCT07154836
Title: Call for Life: Exploring mHealth Solutions for Enhancing Childhood Vaccinations Among Displaced Children in Conflict-affected Settings of Nigeria
Acronym: Call 4 Life
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cambridge (Other)
Collaborators: University of Maiduguri (Other); Infectious Disease Institute at Makerere University (Unknown)
Responsible Party: Principal Investigator, Lundi-Anne Omam Ngo Bibaa, Dr, University of Cambridge
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Call-4-Life; Not application (Other: Cambridge Africa)
Record Dates: First submitted 2025-08-15; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Access to Immunization
Keywords: Immunization; mhealth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Call4life (Experimental): Care givers will be reminded using telephone calls to go vaccine their children
  Interventions: Other: Telephone calls

INTERVENTIONS:
Other: Telephone calls — Regular telephone reminders and health information will be sent to help mothers or caregivers of children 0-23 months to remind them to go vaccine their children
  Other Names: Call4life

SUMMARY:
This study evaluates the feasibility and preliminary impact of Call for Life, an mHealth platform aimed at increasing childhood vaccination coverage among internally displaced persons in Borno State, Nigeria. The platform uses an interactive voice response (IVR) system to deliver automated vaccination reminders, follow up on reported side effects, and provide health messages in English and local languages. A mixed-methods design is used to assess feasibility, interaction rates, and early effects on vaccine uptake. Findings will inform policymakers and humanitarian actors on the potential of mobile technology to strengthen immunization delivery in conflict-affected, resource-limited settings.

ELIGIBILITY:
Inclusion Criteria:

* • Caregivers (male/female) of children from 0-23 months of age or pregnant women in third trimester

  * Caregivers above the age of 18 years of age
  * Caregivers who consent to participate in the study.
  * Resident in the IDP camp for at least one year

Exclusion Criteria:

* • Pregnant women in third trimester in first pregnancy (primigravida)

  * Caregivers that are temporary residents of the IDP camps (IDPs on transit or visitors)
  * Caregivers without the mental capacity to comprehend the questions asked.
  * Inability to use or interact with a mobile phone ( e.g. those with hearing defects or poor vision)

Ages: 23 Months to 23 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 366 (Estimated)
Dates: Start 2025-06-24 (Actual); Primary Completion 2025-11-24 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of zero-dose children aged 0-23 months vaccinated and registered in an immunization registry at the health facility | 6 months
  Number of zero-dose children aged 0-23 months vaccinated and registered in an immunization registry at the health facility. The immunization registry which will be used by the health facility to follow up with parents for the vaccination schedules of the children
Number of care givers to children aged 0-23 months who receive reminder calls from the call for life platform and take their children to the health facility for immunization | 6 months
  Number of care givers to children aged 0-23 months who receive reminder calls from the call for life platform and take their children to the health facility for immunization and registration into an immunization registry

CONTACTS AND LOCATIONS:
Locations (1):
- El Miskin, Jere, Borno State, Nigeria

IPD SHARING:
Plan to Share IPD: Yes
IDP will be shared with researchers involved in the study.
Supporting Information: Study Protocol, SAP
Time Frame: January 2025 to December 2025
Access Criteria: Only researchers involved in the study will have access to IPD